CLINICAL TRIAL: NCT02862054
Title: Splenectomy as a Treatment for Patient With Relapsed Haemophagocytic Lymphohistiocytosis of Unknown Etiology
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Doctor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Splenectomy-HLH
Record Dates: First submitted 2016-08-06; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: haemophagocytic lymphohistiocytosis; splenectomy; unknown etiology
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Splenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Splenectomy (Experimental): Splenectomy as a treatment for patient with relapsed haemophagocytic lymphohistiocytosis of unknown etiology
  Interventions: Procedure: splenectomy

INTERVENTIONS:
Procedure: splenectomy

SUMMARY:
To evaluate the clinical value of splenectomy as a treatment for relapsed haemophagocytic lymphohistiocytosis (HLH) in patient with unknown etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were older than 14 years of age
2. Diagnosed as Hemophagocytic Lymphohistiocytosis (HLH) according to HLH-2004.
3. patients were excluded with infection, rheumatic and immunologic diseases, malignant tumors (especially lymphoma), and primary HLH.
4. Informed consent

Exclusion Criteria:

1. Pregnancy or lactating Women
2. Active bleeding of the internal organs
3. Uncontrollable infection
4. Contraindication of splenectomy
5. Participate in other clinical research at the same time

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | Change from before and1,2,4,8,12 and 24 weeks after splenectomy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.

SECONDARY OUTCOMES:
Survival | from the time patients received splenectomy up to 24 months or December 2018
Adverse events that are related to treatment | through study completion, an average of 2 years
  Adverse events including infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Overall Officials: zhao wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Jing-Shi W, Yi-Ni W, Lin W, Zhao W. Splenectomy as a treatment for adults with relapsed hemophagocytic lymphohistiocytosis of unknown cause. Ann Hematol. 2015 May;94(5):753-60. doi: 10.1007/s00277-014-2276-9. Epub 2014 Dec 16. PMID 25512183